CLINICAL TRIAL: NCT01731561
Title: MAINtenance of Remission Using RITuximab in Systemic ANCA-associated Vasculitis II
Brief Title: Comparison Study of Two Rituximab Regimens in the Remission of ANCA Associated Vasculitis
Acronym: MAINRITSAN 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110146; 2012-001963-66 (EudraCT Number)
Record Dates: First submitted 2012-10-12; First posted 2012-11-22 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis; Renal Limited Forms
Keywords: Granulomatosis with Polyangiitis; Microscopic polyangiitis; Renal limited forms; ANCA-associated vasculitis; Rituximab
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rituximab infusion according biological parameters (Experimental): Rituximab infusion based on ANCA and CD19 lymphocytes
  Interventions: Drug: Rituximab (Arm B)
- Systematic rituximab infusion (Active Comparator): Semestrial rituximab infusion until 18 months
  Interventions: Drug: Rituximab (Arm A)

INTERVENTIONS:
Drug: Rituximab (Arm B) — Rituximab infusion will be performed at D1 then ANCA status and CD19+ lymphocyte count will be monitored every 3 months, and patients will receive new 500 mg rituximab infusions either if CD19 are > to 0/mm3, or if ANCA are positive again or if ANCA titer significantly raises. All patients received corticosteroids, starting from induction with prednisone (or equivalent) at a dose of 1 mg/kg/day with gradual tapering according to a regimen adjusted to body weight over a mean of 18 months since diagnosis.
  Arms: Rituximab infusion according biological parameters
Drug: Rituximab (Arm A) — Rituximab infusion will be performed at D1, D15, M6, M12 and M18(i.e. a total of 5 infusions), at the dose of 500 mg at a fixed dosage.All patients received corticosteroids, starting from induction with prednisone (or equivalent) at a dose of 1 mg/kg/day with gradual tapering according to a regimen adjusted to body weight over a mean of 18 months since diagnosis.
  Arms: Systematic rituximab infusion

SUMMARY:
The aim of this study is to assess the efficacy of a rituximab regimen based on rate of ANCA and CD19 lymphocytes for maintenance treatment in systemic ANCA-associated vasculitis: prospective, multicenter, controlled, randomized comparative study of two rituximab regimens: one based on ANCA and CD19 lymphocytes versus systematic infusions.

DETAILED DESCRIPTION:
Randomized, controlled, national, multicenter, prospective study to compare systematic rituximab infusions (conventional therapy) to rituximab infusion based on rate of ANCA and CD19 lymphocytes in patients with systemic ANCA-associated vasculitis, in remission (achieved with an induction treatment combining corticosteroids and an immunosuppressant after the first flare of the disease (new diagnosis) or after a relapse. Patients will be stratified by first flare (66% of the patients) or relapse (33% of the patients). Patients complying with the inclusion criteria may be included when they are in remission from their vasculitis. Patients will be included at the time of remission and then randomized. They will receive maintenance treatment by 1)2 rituximab infusions mg at D1, D15 then every 6 months until month 18 (i.e. a total of 5 infusions), at the dose of 500 mg. 2) 1 rituximab infusion at the dose of 500 mg at D0 then ANCA status and CD19+ lymphocyte count will be monitored every 3 months, and patients will receive new 500 mg rituximab infusions either if CD19 are > to 0/mm3, or if ANCA are positive again or if ANCA titer significantly raises. After the 18 month length of maintenance phase, i.e. after stopping immunosuppressive maintenance therapy, patients will be followed for an additional 10 month period. Patients with granulomatosis with polyangiitis will be prescribed cotrimoxazole 160/800 tid (for 2 additional years).

ELIGIBILITY:
Inclusion Criteria:

* Granulomatosis with Polyangiitis Or microscopic polyangiitis complying Or kidney-limited disease With or without detectable ANCA (anti-neutrophil cytoplasmic antibodies) at the time of diagnosis or relapse, and at remission.
* Who have achieved remission using a treatment combining corticosteroids and an immunosuppressive agent, including corticosteroids, cyclophosphamide IV or oral (the use of another immunosuppressant is allowed, according to the current French guidelines, as well as plasma exchanges and/or IV immunoglobulins, or rituximab).
* Interval of 1 month between the end of the immunosuppressant treatment and the randomization time if cyclophosphamide or methotrexate were used, interval between 4 and 6 months if rituximab was used
* Age > 18 years without age limit higher when the diagnosis is confirmed.
* Informed and having signed the consent form to take part in the study.

Exclusion Criteria:

* Other systemic vasculitis
* Secondary vasculitis (following neoplastic disease or an infection in particular)
* Induction treatment with a regimen not corresponding to that recommended in France.
* Patient who has not achieved remission.
* Incapacity or refusal to understand or sign the informed consent form.
* Incapacity or refusal to adhere to treatment or perform the follow-up examinations required by the study. Non-compliance
* Allergy, documented hypersensitivity or contraindication to the study medication (cyclophosphamide, corticosteroids, azathioprine, rituximab)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
* Pregnancy, breastfeeding. Women of childbearing age must use a reliable method of contraception throughout the duration of immunosuppressive treatment up to 1 year after the last infusion of rituximab
* Infection by HIV, HCV or HBV
* Progressive, uncontrolled infection requiring a prolonged treatment (tuberculosis, HIV infection, etc.).
* Severe infection declared during the 3 months before randomization (CMV, HBV, HHV8, HCV, HIV, tuberculosis).
* Progressive cancer or malignant blood disease diagnosed during the 5 years before the diagnosis of vasculitis. Patients suffering from non-metastatic prostate cancer or those cured of a cancer or a malignant blood disorder for more than 5 years and not taking any antineoplastic agents for more than 5 years may be included.
* Participation in another clinical research protocol during the 4 weeks before inclusion.
* Any medical or psychiatric disorder which, in the investigator's opinion, may prevent the administration of treatment and patient follow-up according to the protocol, and/or which may expose the patient to a too greater risk of an adverse effect.
* No social security
* Churg and Strauss syndrome
* Viral, bacterial or fungic or mycobacterial infection uncontrolled in the 4 weeks before the inclusion
* History of deep tissue infection (fasciitis, osteomyelitis, septic arthritis)in the first year before the inclusion
* History of chronic and severe or recurrent infection or history of preexisting disease predisposing to severe infection
* Severe immunodepression
* Administration of live vaccine in the four weeks before inclusion
* Severe chronic obstructive pulmonary diseases (VEMS < 50 % or dyspnea grade III)
* Chronic heart failure stade III and IV (NYHA)
* History of recent acute coronary syndrome, unrelated to vasculitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2016-04-05 (Actual)

PRIMARY OUTCOMES:
Number of relapses | at 28 months
  Number of relapses (BVAS>0) majors and minors in each group at the end of the maintenance treatment (18 months treatment + 10 months follow-up)

SECONDARY OUTCOMES:
Number of patients with ANCA (Anti-Neutrophil Cytoplasmatic Antibodies) | at 28 months
  Number of patients with ANCA in each group
Number of adverse events | at 28 months
  To assess the number of adverse events and their severity in each group
Mortality rate | at 28 months
  To assess mortality rate in each group
Number of minor relapse | at 28 months
  number of minor relapse in each group
Cumulated dose of corticosteroid treatment | at 28 months
  Cumulated dose of corticosteroid treatment in each group at 28 months
Number and severity of damages | at 28 months
  Number and severity of damages in each group
Evolution of ANCA and the link of the clinical events | at 28 months
  Evolution of ANCA in each group and the link of the clinical events
Distribution of events by severity | at 28 months
  Distribution of events by severity and it will be assigned to the drug and its mode of administration and/or the severity of the disease (in each group).
Length of corticosteroid treatment | at 28 months
  The length of corticosteroid treatment in each group at 28 months
Rate of B-Lymphocytes CD-19 and the link of the clinical events | at 28 months
  The rate of B-Lymphocytes CD-19 and the link of the clinical events
Evolution of gammaglobulins | at 28 months
Quality of life : SF36 (The Short Form (36) Health Survey) | at 28 months
Functional capacities : HAQ (Health Assessment Questionnaire) | at 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Loic Guillevin, MD, PhD, Study Chair — Cochin Hospital, Paris, France; Pierre Charles, MD, Study Chair — Institut mutualiste, Paris, France
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Background] Charles P, Terrier B, Perrodeau E, Cohen P, Faguer S, Huart A, Hamidou M, Agard C, Bonnotte B, Samson M, Karras A, Jourde-Chiche N, Lifermann F, Gobert P, Hanrotel-Saliou C, Godmer P, Martin-Silva N, Pugnet G, Matignon M, Aumaitre O, Viallard JF, Maurier F, Meaux-Ruault N, Riviere S, Sibilia J, Puechal X, Ravaud P, Mouthon L, Guillevin L; French Vasculitis Study Group. Comparison of individually tailored versus fixed-schedule rituximab regimen to maintain ANCA-associated vasculitis remission: results of a multicentre, randomised controlled, phase III trial (MAINRITSAN2). Ann Rheum Dis. 2018 Aug;77(8):1143-1149. doi: 10.1136/annrheumdis-2017-212878. Epub 2018 Apr 25. PMID 29695500
- [Derived] Khoudour N, Delestre F, Jabot-Hanin F, Jouinot A, Nectoux J, Letouneur F, Izac B, Vidal M, Guillevin L, Puechal X, Charles P, Terrier B, Blanchet B. Association Between Plasma Rituximab Concentration and the Risk of Major Relapse in Antineutrophil Cytoplasmic Antibody-Associated Vasculitides During Rituximab Maintenance Therapy. Arthritis Rheumatol. 2023 Nov;75(11):2003-2013. doi: 10.1002/art.42556. Epub 2023 Aug 13. PMID 37134130
- See also: Website of the French Vasculitis Study Group — http://www.vascularites.org